CLINICAL TRIAL: NCT04224012
Title: Effect of Exercise and Respiratory Therapy on Right Ventricular Function in Severe Pulmonary Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Ekkehard Gruenig, Prof. Dr. med. Ekkehard Grünig; Head of centre for pulmonary hypertension, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TRAIN-01
Record Dates: First submitted 2019-12-19; First posted 2020-01-13 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Exercise; Respiratory Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional therapy group (control group) (No Intervention): patients of the control Group receive usual care
- Interventional group (training group) (Experimental): Specialized exercise and respiratory therapy for patients with pulmonary hypertension
  Interventions: Other: Exercise and respiratory therapy

INTERVENTIONS:
Other: Exercise and respiratory therapy — Three weeks in-Hospital Rehabilitation program with continuation of exercise Training at home
  Arms: Interventional group (training group)

SUMMARY:
Chronic pulmonary hypertension (PH) is associated with impaired exercise capacity, quality of life and right ventricular function.The disease is characterized by an increase of pulmonary vascular resistance and pulmonary arterial pressure, leading to right heart insufficiency. In later stages of the disease, the right heart is not able to further increase right ventricular contractility (cardiac index) during exercise. Within the last decade, new disease-targeted medical therapies have been approved for treatment of pulmonary arterial hypertension (PAH). Sequential and upfront combinations of these agents have shown to further improve symptoms, 6-minute walking distance (6-MWD) and hemodynamics in PAH patients.

Previous training studies have suggested that exercise training as add-on to medical treatment is highly effective improving exercise capacity, quality of life and symptoms. Prospective studies with a 24±12 months follow-up period suggested that exercise training may also improve the rate of clinical worsening events as the need for hospitalization, additional PH-medication, lung-transplantation and death.

There is also first data that exercise training may have a positive impact on the right ventricular function.

This randomised controlled study aims to assess whether exercise training

DETAILED DESCRIPTION:
The aim of this prospective, randomized, controlled study in patients with pulmonary hypertension, who are under stable optimized treatment for at least 2 months, is to examine the effect of an additional exercise and respiratory therapy on the right heart function.

The primary endpoint of this study is the right heart function, measured by cardiac index during exercise invasively determined by right heart catheterization. More hemodynamic parameters for the determination of the right heart function as well as clinical and molecular parameters are relevant to record the physiological effect of the training. The molecular parameters are composed of laboratory parameter and inflammatory parameter as well as genetic analyses, measurements of epigenetic changes measured by microRNA Expressions and DNA-methylation and imunohistochemical measurements of the quadriceps musculature.

The study parameters will be assessed in the patient's routine examinations. Clinical parameters comprise of hemodynamic assessment of pulmonary arterial pressure during exercise, pump function of left and right ventricle, and further echocardiographic parameters. Improvement of exercise capacity will be measured by the change of six-minute walking distance, the breathing economics, the world health organization functional class (WHO functional class), peak oxygen consumption and blood gas analysis. The quality of life will be assessedwith the SF-36 questionnaire.Data for survival analysis will be gained by structured phone interviews . The safety of the training is warranted by long-term, rest- and stress-ECG, safety laboratory, systemic blood pressure, heart frequency, oxygen saturation and occurrence of adverse events. In addition to the routine examinations at baseline and after 15 weeks, a right heart catheterization will be performed.

Patients will be examined in the Thoraxklinik Heidelberg. Patients of the training group will take part in a specific, 3-week inpatient training program at the rehabilitation center Königstuhl Heidelberg right after the baseline examination. The training program consists of exercise and respiratory therapy as well as a mental gait training. Respiratory therapy will be performed 5 times/week for 30 minutes. Furthermore, 15-25 minutes low dosed interval training on a bicycle ergometer, dumbbell training of particular muscle groups with low weights and supervised walks on ground-level will be scheduled 5-7 times/week. Three- to five times a week a "mental gait training" is conducted to estimate the patient's individual physical abilities and limitations. The heart rate during exerciseand the intensity of the training will be closely monitored and individually adjusted. After three weeks of in-hospital rehabilitation the patients are asked to continue the training for twelve further weeks at home. All patients will be examined before the training program, at the end of the in-hospital phase after three weeks and after 15 weeks. Patients of the control group will continue with their lifestyle without individual training prescriptions. After having participated in the study, patients of the control group will also be offered to take part in the training program.

The control examinations cover the medical history, WHO functional class, physical examination, ECG, echocardiography at rest and during exercise, spiroergometry, quality of life, blood-gas analysis, lung function, 6-minute walking distance, oxygen saturation, blood pressure and heart rate, laboratory tests. An optional magnet resonance imaging at the beginning and after three months may also be conducted. At baseline, an optional genetic assessment will be performed; and at the beginning, after three and 15 weeks the expression levels of micro RNA and methylation of the DNA will be assessed. A biopsy of the quadriceps musculature will optionally be carried out at baseline and after 15 weeks. Medication will remain stable throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Consent form
* Men and women >18 years
* Symptomatic PH (WHO-FC II-IV) invasive diagnostis with right heart catheterization: mPAP >25mmHg and a stable optimized treatment for at least 2 month
* Ptients who are able to understand and agree to participate in the study

Exclusion Criteria:

* Pregnancy or breast feeding
* Variation in the medication during the last 2 months
* Patients with signs of right heart decompensation
* Major walking problems
* Unclear diagnosis
* No invasive clarification of the PH
* Acute illness, infections and fever
* Grave lung disease with FEV1 <50% or TLC <70% from target
* Further conclusion criteria are followed: acrive myokarditis, unstable angina pectoris, movement induced venr´tricular rhythmdisturbance, decompensation of the right hart insufficiency, meaningful heartvitien, hyperthrophic obstructive cardiomyopathie or a high grade reduced left ventricular pumpu function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2015-08; Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Cardiac index during exercise, right heart catheter | Change form baseline to final assessment after 15 weeks
  measured by right heart catheterisation; Training vs. control group

SECONDARY OUTCOMES:
Cardiac index at rest, right heart catheter | Change form baseline to final assessment after 15 weeks
  right heart catheterization cardiac index at rest
Pulmonary vascular resistance at rest, right heart catheter | Change form baseline to final assessment after 15 weeks
  right heart catheterization pulmonary vascular resistance at rest
6-minute Walking distance | Change form baseline to final assessment after 15 weeks
  Physical exercise capacity, Walking distance in metres
Peak oxygen consumption, cardiopulmonary exercise testing | Change form baseline to final assessment after 15 weeks
  cardiopulmonary exercise testing
Peak Workload in Watts, achieved during cardiopulmonary exercise testing | Change form baseline to final assessment after 15 weeks
  cardiopulmonary exercise testing
Peak respiratory equivalent during cardiopulmonary exercise testing | Change form baseline to final assessment after 15 weeks
  cardiopulmonary exercise testing
Epigenetic changes of micro RNA | Change form baseline to final assessment after 15 weeks
  Epigenetic changes of the microRNA and the state of methylization (muscle biopsy of the quadrizeps muscuation and peripheral blood)
right atrial area, assessed by echocardiography | Change form baseline to final assessment after 15 weeks
  Echocardiography
right ventricular area, assessed by echocardiography | Change form baseline to final assessment after 15 weeks
  Echocardiography
right ventricular pump function, qualitative during echocardiography | Change form baseline to final assessment after 15 weeks
  Echocardiography
tricuspid annular plane systolic excursion, echocardiography | Change form baseline to final assessment after 15 weeks
  Echocardiography
Physical Summation score, SF-36 | Change form baseline to final assessment after 15 weeks
  Quality of life by short form health Survey 36 (SF-36); values from 0-100 (higher value = better outcome)
Mental Summation score, SF-36 | Change form baseline to final assessment after 15 weeks
  Quality of life by short form health Survey 36 (SF-36)values from 0-100 (higher value = better outcome)
World Health Organization functional class | Change form baseline to final assessment after 15 weeks
  symptoms of pulmonary hypertension
Laboratory: Levels of N-terminal pro brain natriuretic peptide (NT-proBNP) | Change form baseline to final assessment after 15 weeks
  marker of the right heart strain
Oxygen Saturation, blood gas analysis | Change form baseline to final assessment after 15 weeks
  Blood gas analysis
Right heart size, assessed by magnetic resonance tomography | Change form baseline to final assessment after 15 weeks
  magnetic resonance tomography
Right heart function, qualitative, assessed by magnetic resonance tomography | Change form baseline to final assessment after 15 weeks
  magnetic resonance tomography
Clinical worsening, frequency of clinical worsening and adverse Events during the study period | assessed form baseline to final assessment after 15 weeks
  frequency of clinical worsening events

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Pulmonary Hypertension at the Thoraxklinik, Heidelberg University Hospital, Heidelberg, Germany